CLINICAL TRIAL: NCT00404456
Title: The Efficacy of Melatonin in Sleep Problems of Hemodialysis and Peritoneal Dialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meander Medical Center (Other)
Collaborators: Dutch Kidney Foundation (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EMSCAP
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Hemodialysis; Peritoneal Dialysis; Sleep Problems
MeSH Terms: conditions — Parasomnias | interventions — Melatonin

INTERVENTIONS:
Drug: Melatonin — Melatonin 3 mg once-daily

SUMMARY:
Sleep problems can lead to a bad quality of life and a raise of morbidity, also in dialysis patients. Sleep problems can be caused by a disturbance of circadian rhythms in our body. For a good regulation of these circadian rhythms a uniform external synchronisation is necessary. This is the synchronisation of the biological clock of our body by light and other influences. In case of a disturbance of the external synchronisation, due to for example naps during the day or wake periods at night, internal rhythms can be unlinked. As a result a weakened melatonin rhythm and a problematic sleep-wake cycle can be observed. Most dialysis patients have sleep problems. Their sleep latency is prolonged. They often take a nap during the day and their sleep efficiency is poor. There has only been one study on the melatonin rhythm of dialysis patients. The conclusion of this study was that the melatonin rhythm of dialysis patients is weakened and disturbed, probably caused by renal insufficiency. In this study no link was made between melatonin rhythm and the nature and severity of possible sleep problems. In different studies with non-dialysis patients and a disturbed melatonin rhythm, exogenous melatonin at the right time leads to a recovery of the normal rhythm and the normal biological clock and a better quality of life.

The aim is to research the endogenous melatonin rhythm and to improve sleep problems of hemodialysis patients with a placebo-controlled study with exogenous melatonin. Next to this a substudy is performed, in which the effect of the change of daytime to nocturnal in hospital hemodialysis on sleep and melatonin is researched.

ELIGIBILITY:
Inclusion Criteria:

* Stable Peritoneal dialysis
* Stable Hemodialysis
* Age 18-85 years

Exclusion Criteria:

* use of hypnotics, MAO inhibitors or neuroleptics
* Liver disease
* Participation in drug investigation < 1 months to start
* Former use of melatonin
* Severe neurological/psychiatric disease
* Allergic to melatonin or additives

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-04; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Sleep onset latency < 15 minutes
sleep efficiency > 85%
Normalized melatonin rhythm. Dim Light Melatonin Onset (DLMO) 21:00-23:00 hour

CONTACTS AND LOCATIONS:
Overall Officials: Piet ter Wee, MD, PhD, Study Chair — Amsterdam UMC, location VUmc
Locations (1):
- Meander Medical Center, Amersfoort, Netherlands

REFERENCES:
- [Derived] Koch BC, Nagtegaal JE, Hagen EC, van der Westerlaken MM, Boringa JB, Kerkhof GA, Ter Wee PM. The effects of melatonin on sleep-wake rhythm of daytime haemodialysis patients: a randomized, placebo-controlled, cross-over study (EMSCAP study). Br J Clin Pharmacol. 2009 Jan;67(1):68-75. doi: 10.1111/j.1365-2125.2008.03320.x. Epub 2008 Nov 17. PMID 19076157